CLINICAL TRIAL: NCT02488382
Title: Lonquek (Lipegfilgrastim) for Stem Cell Mobilization of Autologous Hematopoietic Stem Cell Transplantation in Patients With Multiple Myeloma and Lymphoma
Brief Title: Lonquek for Autologous Stem Cell Mobilization
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1852-AN-CTIL
Record Dates: First submitted 2015-05-20; First posted 2015-07-02 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma; Multiple Myeloma
Keywords: lymphoma; multiple myeloma; stem cell mobilization; autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lonquek (Experimental): treatment with Lonquek for autologous stem cell collection
  Interventions: Drug: Lonquek

INTERVENTIONS:
Drug: Lonquek — Patients will be given a single fixed dose of Lonquek (Teva LTD), 12-mg subcutaneously.
  Other Names: Lipegfilgrastim

SUMMARY:
The aim of this study is to evaluate the efficacy and tolerability of Lonquek which is a pegylated (long-acting) version of Filgrastim recombinant human G-CSF (G-CSF) in mobilizing sufficient number of stem cells for autologous stem cell transplantation in patients with lymphoma and multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed multiple myeloma or Hodgkins or non Hodgkin lymphoma at need of autologous stem cell transplantation.
* Disease must be chemosensitive or stable status to prior therapy before transplant.
* Age between 18 and 65 years inclusive.
* ECOG performance status 0, 1 or 2.
* Written informed consent.
* Adequate birth control in fertile patients.

Exclusion Criteria:

* Lymphoma patients that did not fulfill the inclusion criteria.
* Patients with factors predicting poor mobilization including >3 lines of previous chemotherapy, extensive irradiation, patients that received stem cell toxicity drugs like Melphalan, Fludarabine, >2 courses of Revlimid, age >65 years, platelets counts <100x109/L, WBC<2.5x109/L or WBC > 35x109/L.
* Previous autologous stem cell transplantation.
* Inability to tolerate peripheral blood stem cell harvest.
* Peripheral venous access not possible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Mobilisation success rate | 4 weeks
  Mobilisation success rate is defined as the mobilisation of a peripheral blood stem cell graft containing >2x106 CD34+ cells/kg in ≤ 4 apheresis sessions.

SECONDARY OUTCOMES:
engraftment after transplantation | 100 days
  Time until recovery of blood counts after transplantation
Safety | 100 days
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Danylesko I, Sareli R, Varda-Bloom N, Yerushalmi R, Shem-Tov N, Magen H, Shimoni A, Nagler A. Long-acting granulocyte colony-stimulating factor pegfilgrastim (lipegfilgrastim) for stem cell mobilization in multiple myeloma patients undergoing autologous stem cell transplantation. Int J Hematol. 2021 Sep;114(3):363-372. doi: 10.1007/s12185-021-03177-9. Epub 2021 Jul 2. PMID 34213732